CLINICAL TRIAL: NCT05003869
Title: Clinical and Basic Research on the Necessity of Scar Tissue Resection During Intrauterine Adhesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lili Cao (Other)
Responsible Party: Sponsor-Investigator, Lili Cao, Shandong Qianfoshan Hospital Scientific Research Department Director, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QCT042806
Record Dates: First submitted 2021-07-14; First posted 2021-08-13 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Intrauterine Adhesion; Scar
MeSH Terms: conditions — Gynatresia; Cicatrix

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoperative resection of intrauterine scar tissue by TCRA (Experimental): Study group: patients took the bladder lithotomy position, routinely disinfected vulva and vagina, and laid sterile towel and sheet.pliers Clamp the front lip of the cervix, explore the depth of the uterine cavity, dilate the cervical canal one by one, place the endoscopy, and examine the uterine cavity.After the scar tissue contracted on one side, the scar tissue was disintegrated at the boundary between the intima and scar tissue. The scar tissue was removed with the annular electrode, and a balloon was placed after surgery to prevent re-adhesion.Complete adhesion release is defined as a return to normal shape of the uterine cavity with bilateral uterine angles exposed.
  Interventions: Procedure: Scar tissue is removed
- No scar tissue resection group (No Intervention): During the operation, the scar tissue covering the anterior, posterior and lateral walls of the uterine cavity was ploughed longitudinally into several narrow strips with needle-like electrodes, and scar tissue was not excised.

INTERVENTIONS:
Procedure: Scar tissue is removed — The patients were divided into two groups according to whether the scar tissue was removed during TCRA operation: study group: resection of uterine scar tissue during TCRA operation;In the control group, the scar tissue covering the anterior, posterior and lateral walls of the uterine cavity was ploughed longitudinally into several narrow strips using needle-like electrodes, and the scar tissue was not excised.
  Other Names: No scar tissue is removed
  Arms: Intraoperative resection of intrauterine scar tissue by TCRA

SUMMARY:
TCRA is an important surgical method to restore normal menstrual cycle and improve the outcome of pregnancy.However, postoperative intrauterine adhesion, uterine cavity deformation and difficulty in normal intimal growth seriously affect the efficacy of surgery. A large number of existing studies have shown that even after surgical treatment, women with a history of IUA are still at a reproductive disadvantage.Whether scar tissue plays a role in these influencing factors? At present, there is a variety of surgical methods, and there is no clear guideline consensus on how to deal with intrauterine scar tissue during surgery.

DETAILED DESCRIPTION:
Intrauterine adhesions (IUA) are pathological symptoms of endometrial basal layer damage, fibrous tissue formation and tissue bridge between uterine walls caused by a variety of reasons.In recent years, with the increase of uterine operations such as hysterotomy and cesarean section, the incidence of IUA has been increasing year by year.IUA is mainly manifested by reduced menstrual volume, amenorrhea, recurrent abortion, infertility and abnormal implantation of embryos, etc., which poses a great threat to the health and quality of life of patients.Transcervieal resection of adhesions (TCRA) is a targeted method to separate intrauterine adhesions under direct vision and basically restore the morphology of the intrauterine cavity. It is an important surgical method to improve the pregnancy outcome.However, a large number of existing studies have shown that women with a history of IUA remain at a reproductive disadvantage even after surgical treatment.

Based on the current situation, the investigators have designed this topic, to conduct a study on TCRA intraoperative scar tissue to remove the necessity of clinical and basic research, explore the scar tissue resection or not for the clinical curative effect and the effect of combined tissue morphology, molecular biology research, for TCRA intraoperative how to deal with the scar tissue provide a certain amount of practice and theory basis.

Estrogen receptor (e-r) and progesterone receptor (P - R) is located in the nucleus, when the receptor and hormones to form complexes, again in the form of activation combined into specific areas of the chromosome, gene activation, synthesis of new DNA transcription, and synthesis of new proteins, through the biological function of protein regulating cell growth and metabolism.Specifically, they participate in the reconstruction and regeneration of endometrial blood vessels and cells.The number and functional status of hormone receptors determine the local levels of estrogen and progesterone that can exert biological effects. If the expression of E-R and P-R is reduced or the function is abnormal, the sensitivity and reactivity of endometrium to hormones will be directly reduced, and the endometrial growth will be affected.

The treatment of IUA is mainly based on direct separation of the adhesive tissue, supplemented by the corresponding hormone or cytokine therapy.Among them, estrogen is widely used.On the one hand, it plays a corresponding role by binding with receptors; on the other hand, it affects the fibrinogen and extracellular matrix deposition by regulating the expression of TGF-β or MMP-9, thus participating in the occurrence of intrauterine adhesions.

Studies have found that there is a certain correlation between transforming growth factor-β1 (TGF-β1) and the pathogenesis of IUA. TGF-β1 is a kind of cytokine that is synthesized and secreted by lymphocytes, macrophages, platelets and other cells and can regulate cell growth and differentiation, belonging to the TGF family.It can promote tissue fibrosis and extracellular matrix production, and can increase the amount of fibronectin and collagen.However, a number of studies have confirmed that inhibiting the expression of TGF-β1 or reducing its activity can effectively reduce the degree of fibrosis in liver, kidney and other tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Consensus of Chinese Experts on the Clinical Diagnosis and Treatment of Intrauterine Adhesions, i.e., patients with previous history of induced abortion and other intrauterine operations, accompanied by periodical abdominal pain, fewmenorrhea, amenorrhea, recurrent abortion, infertility, and uterine adhesions found by hysteroscopy, who have fertility requirements;
2. According to the American Reproductive Society prognostic classification, the AFS score was moderate to severe intrauterine adhesions, that is, the score range was 5-12 points;
3. Patients ranged in age from 18 to 42 years old;
4. normal endocrine function and ovulation;
5. Patients had comprehensive clinical data and were followed up after surgery.

Exclusion Criteria:

1. Patients with severe cardiovascular and cerebrovascular diseases, liver and kidney dysfunction and other systemic diseases;
2. Patients who recently received female genital surgery or underwent high uterine flexion and were unable to receive hysteroscopy and surgical treatment;
3. Amenorrhea, recurrent abortion and infertility caused by other factors such as neuro-endocrine system disorders or congenital abnormalities of reproductive structure and development;
4. Patients with allergic reaction to estrogen and other drugs;
5. Severe abnormal semen of the spouse.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
The menstrual chart records changes in menstrual volume | 1 to 3 months before surgery and the first month after the operation
  Menstrual chart records the amount of menstruation before and after surgery:Menstrual volume is basically normal;Menstrual volume increased compared with preoperative;Still amenorrhea or menstrual volume is not increased
Preoperative and postoperative changes in endometrial thickness were recorded by Doppler ultrasonography. | Ultrasound examinations were performed before and 2 weeks after the first operation, and 2 weeks after the second operation
  Ultrasound was used to record endometrial thickness before and 2 weeks after the first operation. The second hysteroscopy was performed 3-7 days after the first clean menstruation after the first operation, and ultrasound was performed again 2 weeks after the operation to record the data and compare the endometrial thickness of each group.
Preoperative and postoperative changes of intrauterine adhesions were recorded according to the American Fertility Society score in 1988: mild :1 ~ 4; Moderate: 5-8; Severe: 9-12 points | The first operation time is 3-7 days after menstruation (excluding amenorrhea pregnancy can be operated at any time). The second operation was performed 1 month after the first operation
  The operation time was within 3-7 days after menstruation (surgery could be performed at any time after excluding pregnancy for amenorrhea). Preoperative hysteroscopy scores and surgical procedures were all performed by the same surgeon.Intrauterine adhesions were measured using the 1988 American Fertility Society (AFS) score.
  Three to seven days after the first menstrual cleanness, the patient was admitted to the hospital for hysteroscopic reexamination. During hysteroscopy, the intrauterine adhesion and intimal recovery of the patient were explored.

SECONDARY OUTCOMES:
Ultrasound of uterine adnexa was used to record the intrauterine pregnancy | The pregnancy of the patients was followed up by telephone three months after surgery for at least 1 year, and the clinical pregnancy rate was recorded.
  The pregnancy of the patients was followed up by telephone three months after surgery for at least 1 year, and the clinical pregnancy rate was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yingchun Ma, Doctor, Study Chair — Shandong First Medical University
Locations (1):
- China, Shandong Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Personal data of participants and participants in the study will be kept confidential and will only be used for statistical analysis by the study team